CLINICAL TRIAL: NCT03506178
Title: The Effects of Nasal Airflow on Upper Airway Dilator Muscles During Sleep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: TRECKY2017-1109
Record Dates: First submitted 2018-04-12; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Upper airway; Obstructive sleep apnea; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obstructive sleep apnea patients (Experimental)
  Interventions: Drug: Oxymetazoline Nasal Spray; Drug: Menthol Nasal Spray; Drug: Normal saline Nasal Spray; Device: Nasal mask with partly blocked
- Healthy controls (Other)
  Interventions: Drug: Oxymetazoline Nasal Spray; Drug: Menthol Nasal Spray; Drug: Normal saline Nasal Spray; Device: Nasal mask with partly blocked

INTERVENTIONS:
Drug: Oxymetazoline Nasal Spray — Obstructive sleep apnea (OSA) Patients and healthy controls were treated with 4 different nasal intervention ,including Oxymetazoline Nasal Spray,Normal saline Nasal Spray,Menthol Nasal Spray or Nasal mask with partly blocked when they sleep onset. At the treatment periods, polysomnograpy, genioglossus enlectromyography, pharyngeal current perception threshold and sleep quality scores were assess.
Drug: Menthol Nasal Spray — Obstructive sleep apnea (OSA) Patients and healthy controls were treated with 4 different nasal intervention ,including Oxymetazoline Nasal Spray,Normal saline Nasal Spray,Menthol Nasal Spray or Nasal mask with partly blocked when they sleep onset. At the treatment periods, polysomnograpy, genioglossus enlectromyography, pharyngeal current perception threshold and sleep quality scores were assess.
Drug: Normal saline Nasal Spray — Obstructive sleep apnea (OSA) Patients and healthy controls were treated with 4 different nasal intervention ,including Oxymetazoline Nasal Spray,Normal saline Nasal Spray,Menthol Nasal Spray or Nasal mask with partly blocked when they sleep onset. At the treatment periods, polysomnograpy, genioglossus enlectromyography, pharyngeal current perception threshold and sleep quality scores were assess.
Device: Nasal mask with partly blocked — Obstructive sleep apnea (OSA) Patients and healthy controls were treated with 4 different nasal intervention ,including Oxymetazoline Nasal Spray,Normal saline Nasal Spray,Menthol Nasal Spray or Nasal mask with partly blocked when they sleep onset. At the treatment periods, polysomnograpy, genioglossus enlectromyography, pharyngeal current perception threshold and sleep quality scores were assess.

SUMMARY:
Obstructive sleep apnea (OSA) is an increasingly prevalent disorder characterized by repeated upper airway collapse during sleep, resulting in oxygen desaturation and frequent arousals. The etiology of OSA remains unclear.

Many studies indicates an association between nasal obstruction and apnea. However,the precise nature of this relationship is far from clear and the importance of resistance to nasal airflow in the pathogenesis of airway collapse in OSA patients remains contentious.

In this study, investigators perform 4 different ways to change subjective or objective patency of nasal cavity and observe the effects of the nasal airflow on nocturnal breathing, sleep,and upper airway muscles in OSA patients.

DETAILED DESCRIPTION:
1. All subjects underwent a standard overnight polysomnogram(PSG), including continuous genioglossal electromyography measurement , electroencephalogram, electrooculogram, electrocardiogram, nasal flow (thermister), respiratory (chest and abdominal) movements,oxy-hemoglobin saturation (pulse oximeter), and body position. Apnea event definitions and clinical classification were determined using the American Academy of Sleep Medicine(AASM) guidelines
2. Pharyngeal electrical current sensory threshold was performed to identify the different Pharyngeal function between OSA patients and normal controls

ELIGIBILITY:
Inclusion Criteria:

* OSA patients (apnea/hyponea index >5/h）with chronic nasal congestion

Exclusion Criteria:

* Upper airway surgery;
* Current treatment with nasal topical steroids or decongestants;
* Internal medical diseases or psychiatric disorders that interferd with sleep.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-05-12 (Estimated); Study Completion 2018-05-12 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea Index | 2 to 6 month
  A randomized, placebo-controlled double blind study on the effects of nasal spray oxymetazoline on sleep architecture, respiratory events, body position and subjective scores in OSA patients. All participants received specific physical examinations, subjective scale assessments and a two-night polysomnography sduty (by randomly applying oxymetazoline for one night and placebo for another.).Data collected after oxymetazoline or placebo treatments were compared. Apnea-hypopnea index(AHI),defined as the sum of apneas and hypopneas per sleep hour, was used as an important indicator for assess the severity of OSA.
Myoelectricity of genioglossus | 2 to 6 month
  Participants were treated with 4 different nasal intervention ,including Oxymetazoline Nasal Spray, Normal saline Nasal Spray, Menthol Nasal Spray or Nasal mask with partly blocked when they sleep onset. At the treatment periods, subjects underwent overnight polysomnography with synchronous genioglossus electromyography . Genioglossus (GG) activations under different nasal ventilation conditions were compared.
The pharyngeal current sensory threshold | 2 to 6 month
  The pharyngeal current perception threshold test was performed before and after different nasal intervention including Oxymetazoline Nasal Spray, Normal saline Nasal Spray, Menthol Nasal Spray or Nasal mask with partly blocked different nasal cavities. Data collected from OSA patients and healthy controls were compared and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Demin Han, MD,PhD, Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] An Y, Gao F, Su X, Zhou C, Huang J, Chen S, Liu T, Lu Z. Characteristics of pharyngeal paraesthesia symptoms in patients with obstructive sleep apnoea. Sleep Breath. 2021 Dec;25(4):2163-2169. doi: 10.1007/s11325-021-02325-z. Epub 2021 Feb 18. PMID 33604802
- [Derived] An Y, Li Y, Chang W, Gao F, Ding X, Xu W, Han D. Quantitative Evaluation of the Function of the Sensory Nerve Fibers of the Palate in Patients With Obstructive Sleep Apnea. J Clin Sleep Med. 2019 Sep 15;15(9):1347-1353. doi: 10.5664/jcsm.7756. PMID 31538606
- [Derived] An Y, Li Y, Kang D, Sharama-Adhikari SK, Xu W, Li Y, Han D. The effects of nasal decongestion on obstructive sleep apnoea. Am J Otolaryngol. 2019 Jan-Feb;40(1):52-56. doi: 10.1016/j.amjoto.2018.08.003. Epub 2018 Aug 23. PMID 30243839